CLINICAL TRIAL: NCT06558643
Title: A First-in-Human, Single-Centre, Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of a Single Intramuscular Injection of MMV371 Long-Acting Injection Formulation in Healthy Participants
Brief Title: Single Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of MMV371 LAI in Healthy Participants
Acronym: MV371 LAI FiH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Quotient Sciences (Industry); The Doctors Laboratory Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MMV_MMV371_23_01_FIH
Record Dates: First submitted 2024-07-25; First posted 2024-08-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Malaria,Falciparum
Keywords: Malaria; First in Human; Healthy Volunteers
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: Three cohort, single ascending dose, randomised, double-blinded, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: Appearance matching of the placebo is not possible; therefore, non-blinded dosing teams will be used to preserve the study blind. IMP labels will state MMV371 or placebo and use a common expiry date. IMP accountability logs will be maintained by unblinding the randomisation schedule and disclosure envelopes will be generated by an unblinded statistician. The unblinded statistician will not be involved in any decisions relating to populations for analysis or study decisions prior to unblinding. Documentation and unblinded files will be stored in a secure location and shared with unblinded staff only using sealed envelopes. Interim PK parameter estimations will be performed using bioanalytical data applied with participant aliases. There may be instances where interim PK data have the potential to be treatment revealing. Every effort will be made by the pharmacokineticist to maintain the study blind by appropriate presentation of data to the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 Single Ascending Dose Regime A (Experimental): MMV371 Long-acting injection (LAI) 112mg (0.5 ml) or Placebo for MMV371 Long-acting injection(0.5 ml)
  Interventions: Drug: MMV371 LAI; Drug: Placebo for MMV371
- Cohort 2 Single Ascending Dose Regime B (Experimental): MMV371 Long-acting injection (LAI) 223mg (1.0 ml) or Placebo for MMV371 Long-acting injection (1.0 ml)
  Interventions: Drug: MMV371 LAI; Drug: Placebo for MMV371
- Cohort 3 Single Ascending Dose Regime C (Experimental): MMV371 Long-acting injection (LAI) 446mg (2.0 ml) or Placebo for MMV371 Long-acting injection (2.0 ml)
  Interventions: Drug: MMV371 LAI; Drug: Placebo for MMV371
- Cohort 4 Single Ascending Dose Regime D (Experimental): MMV371 Long-acting injection (LAI) 669mg (3.0 ml) or Placebo for MMV371 Long-acting injection (3.0 ml)
  Interventions: Drug: MMV371 LAI; Drug: Placebo for MMV371

INTERVENTIONS:
Drug: MMV371 LAI — Single intra-muscular dose
Drug: Placebo for MMV371 — Single intramuscular dose

SUMMARY:
This three-cohort, first-in-human, healthy participant study aims to assess the test medicine's safety and tolerability, including injection site reactions and how it is taken up by the body when given as a single dose.

For Cohort 1, up to 8 participants will be randomly assigned to receive the starting dose of the test medicine or dummy medicine (placebo) as a single intramuscular injection.

For Cohort 2, if the safety and tolerability results from Cohort 1 are satisfactory, up to 8 participants will be randomly assigned to receive double the starting dose of the test medicine or dummy medicine (placebo) as a single intramuscular injection.

For Cohort 3, if the safety and tolerability results from Cohort 1 are satisfactory, up to 8 participants will be randomly assigned to receive double the Cohort 2 dose of the test medicine or dummy medicine (placebo) as a single intramuscular injection.

Participants' blood and urine will be taken throughout the study for analysis of the test medicine and for their safety. When in the clinical unit, the injection site will be checked daily for reactions, and a diary will be provided on discharge for further recording. Participants will be discharged 6 days after dosing and return to the clinical unit an additional 9 times for for safety assessments to be performed. Participants are expected to be involved in this study for approximately 12 weeks for all study activities, from screening to the final return visit.

DETAILED DESCRIPTION:
This is a single-centre, participant- and investigator-blind, randomised, placebo-controlled, single ascending dose (SAD) study to assess the safety, tolerability and PK of a single intra-muscular depot injection of MMV371 long-acting injection (LAI) formulation in healthy participants.

It is planned to enrol 3 sequential cohorts of up to 8 healthy male participants and healthy non-pregnant, non-lactating female participants. In each cohort, participants will be randomised in a ratio of 6 active IMP to 2 placebo.

All cohorts will follow a sentinel dosing design. On Day 1, two sentinel participants (sentinel group) will be randomly assigned to receive a single IM dose of either active investigational medicinal product (IMP) or placebo (1 participant each) to assess safety (with a focus on acute severe toxicity) and tolerability, including injection site reactions (ISRs).

The sentinel group will be dosed concomitantly at least 48 h prior to the rest of the cohort (main group). The main group will comprise 6 participants randomly assigned to receive a single IM dose of either active IMP or placebo in a 5:1 ratio to assess safety and tolerability (including ISRs).

An interim data review of the safety, tolerability (including ISRs), and PK data obtained up to Day 15 for each cohort will be conducted prior to the dose decision for the subsequent cohort(s). Should the data suggest that it is safe to proceed to the next dose group, progression to that group will be permitted.

The starting dose will be 112 mg MMV371, and dose escalation between SAD cohorts will be a maximum of 2-fold. No dose selected will exceed 446 mg MMV371.

* Cohort 1 will receive Regime A : MMV371 (112 mg (0.5 mL), or placebo.
* Cohort 2 will receive Regime B: MMV371 (223 mg (1.0 mL), or placebo.
* Cohort 3 will receive Regime C: MMV371 (446 mg (2.0 mL), or placebo.

In each cohort, participants will be dosed on Day 1 and will remain residents in the clinical unit until discharge on Day 6. They will be required to return to the clinical unit on Days 8, 10, 12, 15, 18, 23, 29, and Week 8 for the assessments detailed in the schedule of assessments and Week 12 for the end-of-study assessment.

For all parts, blood samples will be collected at regular intervals for PK analysis and safety from Day 1 to discharge from the study. Participants will also be trained to complete an Injection Site Reaction Diary(ISRD) whilst resident in the clinical unit. They will receive an ISRD at discharge on Day 6 and at each return visit until the EOS visit. The ISRD should be completed at home to document new, changing or re-appearing ISRs on non-visit days/weeks; changes at the injection site or the re-appearance of an ISR(s) should be recorded in the diary whenever they occur.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent
2. Must be willing and able to communicate and participate in the whole study Aged 18 to 64 years inclusive at the time of signing informed consent

4. Must agree to adhere to the contraception requirements defined in Section 9.4 of the Protocol 5. Healthy males or non-pregnant, non-lactating healthy females, determined by normal physical examination, safety bloods, urinalysis, ECG and vital sign assessments 6. Body mass index (BMI) of 19.0 to 32.0 kg/m2 as measured at screening 7. Weight ≥50 kg for males and ≥45 kg for females at screening

Exclusion Criteria:

1. Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients, Wellvone®/Mepron® and/or Malarone®
2. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
3. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
4. Blood pressure (BP; supine) at screening or pre-dose outside the range of 90 to 140 mmHg systolic BP in participants ≤45 years, 90 to 150 mmHg SBP in participants >45 years or 50 to 90 mmHg diastolic BP; and pulse rate outside the range of 45 to 100 bpm, unless deemed not clinically significant by the investigator
5. History or presence of known structural cardiac abnormalities, family history of long QT syndrome, cardiac syncope or recurrent, idiopathic syncope, exercise related clinically significant cardiac events. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QT interval changes
6. Presence of sinus node dysfunction, clinically significant PR interval prolongation (>220 msec), intermittent second- or third-degree atrioventricular block, complete bundle branch block, sustained cardiac arrhythmias including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles, abnormal T wave morphology which may impact on the QT/QTc assessment, or QTcF >450 msec.
7. Participants with a history of cholecystectomy or gall stones.
8. Participants who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
9. Participants with tattoos or scars or other significant dermatological conditions overlying the deltoid region which may interfere with injection site assessments, as determined by the investigator or delegate at screening.
10. Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1). Participants with Gilbert's Syndrome are not allowed
11. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results.
12. Transaminases (ALT or AST) >ULN
13. Females who are pregnant or lactating (all female participants must have a negative highly sensitive serum pregnancy test at screening and a negative urine pregnancy test at admission).
14. Participants who have received any IMP in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
15. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood.
16. Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day, up to 800 mg ibuprofen per day, hormonal contraception or HRT) in the 14 days before IMP administration (see Section 11.4). Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no pharmacodynamic activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardise the safety of the trial participant; and if the use of medication is not considered to interfere with the objectives of the study.
17. Participants who are taking, or who have taken, rifampin/rifabutin, tetracycline and indinavir in the 30 days before IMP administration
18. Participants who have had a COVID-19 vaccine within 14 days before dosing.
19. History of any drug or alcohol abuse in the past 2 years
20. Regular alcohol consumption in males >21 units per week and in females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
21. A confirmed positive alcohol breath test at screening or admission
22. Current smokers and those who have smoked within the last 12 months
23. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
24. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
25. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1) at screening or admission
26. Male participants with pregnant or lactating partners
27. A score of SI 4 to 5 (related to suicidal ideation) or any SB score (related to suicidal behaviour) as assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening.
28. Participants who are, or are immediate family members of, a study site or sponsor employee.
29. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) as assessed by the investigators. | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  AEs (including SAEs),whether ascribed to study procedures or not, will be recorded from the time of providing written informed consent until the EOS visit/unscheduled follow-up visit. Participants will be asked to self-report any new, changing or re-appearing AEs in the 30 days after the Week 12 EOS visit.
  Descriptive summaries of AE assessments by treatment will be provided.
Number of participants with injection site reactions (ISRs) as assessed by DAIDS grading scale v2.1 | Dosing (Day 1) up to 30 days after end of study (EOS) visit.
  At scheduled time points (0.5hr; 1hr; 2hr; 4hr; 6hr; 8hr; 12hr; 24hr; 48hr; 72hr; 96hr; 120hr; 168hr; 216hr; 264hr; 336hr; 408hr; 528hr; 672hr; 1344hr and 2016hr), following IMP administration, the injection site will be examined for presence of the following ISRs, which will be graded from Grade 1 (mild) to Grade 4 (potentially life-threatening), according to the DAIDS grading scale:
  * Injection site pain/tenderness
  * Injection site erythema/redness
  * Injection site induration/swelling
  * Injection site pruritis The presence and/or severity of erythema/redness and induration/swelling at the injection site will be assessed using the largest dimension.
  Participants will be provided with an Injection Site Reaction Reaction Diary (ISRD) on discharge from the unit on Day 6 for recording new, changing, or reappearing ISRs on non-visit days/weeks.
  Any clinically significant ISR will be reported as an AE as per the judgement of the investigator.
Number of participants that present with injection site nodules assessed and recorded using a four-point scale. | Dosing (Day 1) up to 30 days after end of study (EOS) visit.
  At scheduled time points (0.5hr; 1hr; 2hr; 4hr; 6hr; 8hr; 12hr; 24hr; 48hr; 72hr; 96hr; 120hr;168hr; 216hr; 264hr; 336hr; 408hr; 528hr; 672hr; 1344hr and 2016hr), following IMP administration, the injection site will be examined for presence of nodules, which will be scored from 0 (no nodule) to 3 (Large nodule >1cm in diameter).
  Injection Site Nodule Examination Score Nodules 0 No nodule
  1. Small nodule <0.5 cm in diamete4
  2. Medium size nodule 0.5 to 1 cm in diameter
  3. Large nodule >1 cm in diameter
  Participants will receive an Injection Site Reaction Reaction Diary (ISRD) on discharge from the unit on Day 6 for recording new, changing, or reappearing nodules on non-visit days/weeks.
  Any clinically significant ISR will be reported as an AE as per the investigator's judgement.
Number of participants with abnormal findings during targeted Physical examination and/or Adverse Events related to treatment: | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  During the targeted (symptom-driven) physical examination (216hr; 672hr; 1344hr and 2016hr), following IMP administration, a physician will assess the participant; if the participant reports feeling unwell or has ongoing AEs, the physician will examine the appropriate body system(s) if required.
  Examination of lymph nodes (mandibular, axillar and inguinal) for changes such as swelling and hardening (induration) will be conducted.
  Descriptive summaries of physical assessments by treatment will be provided.
Number of participants with abnormal safety blood results and/or Adverse Events related to treatment). | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  Safety blood samples collected at time points (Screening, admission; pre-dose; 4hr; 48hr; 216hr; 408hr; 672hr; 1344hr and 2016hr) are assessed for lab values for (haematology, coagulation (only pre-dose; 4hr; 408hr), biochemistry and urinalysis) that move out of the normal range will be noted and assessed for clinical significance. Any clinically significant abnormality, including changes from baseline, must be reported as an AE.
Number of participants with abnormal electrocardiograms (ECGs) and/or Adverse Events related to treatment). | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  Triplicate ECGs are collected at the following time points (Screening, pre-dose; 4hr; 48hr; 216hr; 408hr; 672hr; 1344hr and 2016hr). The mean value for the triplicate ECGs (supine) will be reviewed for safety assessments. Any clinically significant abnormality, including changes from baseline, will be reported as an AE.
  Absolute QTcF prolongation
  * QTcF >450 msec
  * QTcF >480 msec
  * QTcF >500 msec Change from baseline in QTcF
  * QTcF increases from baseline >30 msec
  * QTcF increases from baseline >60 msec
Number of participants with abnormal vital signs and/or Adverse Events related to treatment: Blood pressure | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  Blood pressure is measured in millimetres of mercury (mmHg), at the following time points (Screening, pre-dose; 4hr; 48hr; 216hr; 408hr; 672hr; 1344hr and 2016hr) with the participant supine for a minimum of 5 minutes.
  Any clinically significant abnormality, including changes from baseline, must be reported as an AE.
Number of participants with abnormal vital signs and/or Adverse Events related to treatment: Heart rate. | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  Heart rate is measured in beats per minute (bpm), at the following time points (Screening, pre-dose; 4hr; 48hr; 216hr; 408hr; 672hr; 1344hr and 2016hr) with the participant supine for a minimum of 5 minutes.
  Any clinically significant abnormality, including changes from baseline, must be reported as an AE.
Number of participants with abnormal vital signs and/or Adverse Events related to treatment:Respiration Rate | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  Respiration rate is measured in breaths per minute at the following time points (Screening, pre-dose; 4hr; 48hr; 216hr; 408hr; 672hr; 1344hr and 2016hr) with the participant supine for a minimum of 5 minutes.
  Any clinically significant abnormality, including changes from baseline, must be reported as an AE.
Number of participants with abnormal vital signs and/or Adverse Events related to treatment: Body temperature. | Screening/Day-28 up to 30 days after end of study (EOS) visit.
  Body temperature is measured in degrees centigrade (°C), at the following time points (Screening, pre-dose; 4hr; 48hr; 216hr; 408hr; 672hr; 1344hr and 2016hr) with the participant supine for a minimum of 5 minutes.
  Any clinically significant abnormality, including changes from baseline, must be reported as an AE.
Participants' Weight in kilograms (kg) | Screening and Admission
  Weight is measured at Screening and Admission and will be combined with Height in centimetres (cm) to report BMI in kg/m^2
Participants' Height in centimetres (cm) | Screening
  Weight is measured at Screening and Admission and will be combined with Height in centimetres (cm) to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, MD, DPM, FFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom